CLINICAL TRIAL: NCT00354276
Title: A Phase II Study of Cloretazine® (VNP40101M) for Elderly Patients With De Novo Poor Risk Acute Myelogenous Leukemia
Brief Title: VNP40101M Followed by Cytarabine in Treating Older Patients With Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vion Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000492755; VION-CLI-043; EUDRACT-2006-001853-89; NCT00389623 (obsolete NCT alias)
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2009-05

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(16;16)(p13;q22); untreated adult acute myeloid leukemia; adult acute myelomonocytic leukemia (M4); adult acute monocytic leukemia (M5b); adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); adult acute monoblastic leukemia (M5a); adult acute megakaryoblastic leukemia (M7); adult acute basophilic leukemia; adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute eosinophilic leukemia; adult acute minimally differentiated myeloid leukemia (M0)
MeSH Terms: conditions — Leukemia; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Basophilic, Acute; Leukemia, Myeloid, Acute; Leukemia, Eosinophilic, Acute | interventions — Cytarabine; laromustine

INTERVENTIONS:
Drug: cytarabine
Drug: laromustine

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as VNP40101M and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving VNP40101M followed by cytarabine may kill more cancer cells.

PURPOSE: This phase II trial is studying how well VNP40101M followed by cytarabine works in treating older patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the complete response rate in older patients with poor-risk, de novo acute myeloid leukemia treated with VNP40101M as induction therapy followed by cytarabine as consolidation therapy.

Secondary

* Determine the probability of overall survival, leukemia-free survival, and progression-free survival of patients treated with this regimen.
* Determine the safety of this regimen in these patients.

OUTLINE: This is an open-label, multicenter study.

* Induction therapy: Patients receive VNP40101M IV over 60 minutes on day 1 (course 1). Patients without evidence of disease progression who have responding but residual disease receive a second course of VNP40101M once between days 35-60. Patients achieving complete response or partial response after induction therapy proceed to consolidation therapy.
* Consolidation therapy: Beginning between days 45-90, patients receive cytarabine IV continuously over 5 days (course 1). Patients may receive a second course of cytarabine at the discretion of the investigator.

After completion of study treatment, patients are followed periodically for up to 36 months.

PROJECTED ACCRUAL: A total of 85 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed de novo acute myeloid leukemia (AML)

  * No acute promyelocytic leukemia [t(15;17)]
  * No favorable cytogenetics, including t(15;17), t(8;21), or inv 16
  * No secondary AML, defined as having a history of an antecedent hematologic disorder (myelodysplastic syndromes [MDS] or myeloproliferative disease), or history of prior chemotherapy or radiation for a disease other than AML
* Must have ≥ 1 of the following poor-risk features:

  * Any of the following unfavorable cytogenetics:

    * Del (5q)/-5q
    * -7/del(7q)
    * Abnormal 3q, 9q, 11q, 20q, 21q, or 17p
    * t(6;9)
    * t(9;22)
    * Trisomy 8
    * Complex karyotypes (≥ 3 unrelated abnormalities)
  * At least 70 years of age
  * ECOG performance status (PS) of 2
  * Cardiac dysfunction* that would limit the use of anthracycline therapy, as defined by any of the following:

    * Ejection fraction ≤ 50%
    * History of significant coronary artery disease, defined as ≥ 1 vessel stenosis requiring medical treatment, stent placement, or surgical bypass graft
    * History of congestive heart failure or myocardial infarction
    * Significant arrhythmia, including any of the following:

      * Atrial flutter (excluding atrial fibrillation)
      * Sick sinus syndrome
      * Ventricular arrhythmia
    * Heart valve disease

      * Mitral valve prolapse allowed
    * Other heart disease, at the discretion of the principal investigator
  * Pulmonary dysfunction not related to AML, defined by 1 of the following:

    * DLCO and/or FEV_1 < 80% and ≥ 50% normal range
    * Dyspnea on slight activity or at rest
    * Requires oxygen
  * Hepatic dysfunction related to chronic hepatitis or liver cirrhosis
  * Other organ dysfunction or comorbidity that precludes standard cytotoxic induction treatment (e.g., "3+7"), at the discretion of the principal investigator NOTE: *Patients with a history of heart disease as defined above must be on appropriate medication and have their disease under control
* No known CNS disease

PATIENT CHARACTERISTICS:

* ECOG PS 0-2
* AST and ALT ≤ 5 times upper limit of normal
* Bilirubin ≤ 2.0 mg/dL
* Creatinine ≤ 2.0 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after completion of study treatment
* No active, uncontrolled infection

  * Patients with an infection who are under active treatment with antibiotics and whose infections are controlled are eligible
  * Chronic hepatitis allowed
* No clinical evidence of ongoing second malignancy unrelated to AML or MDS
* No evidence of left bundle branch block on screening ECG
* No obligate use of cardiac pacemaker or atrial fibrillation

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 24 hours since prior metronidazole
* No prior low-dose, single-agent, cytotoxic chemotherapy (e.g., cytarabine, decitabine, or azacitidine)
* No concurrent disulfiram
* No other concurrent standard or investigational therapy for AML except for the following:

  * Concurrent hydroxyurea to control rising white blood cell counts

    * Dosage must be 4-6 grams daily for up to 4 days
  * Concurrent leukapheresis to control blast cell counts

    * Must be completed within the first 5 days of study therapy
    * No more than 2 procedures per day or 4 procedures total
  * Investigational supportive care agents (e.g., antimicrobials or antifungal agents), at the discretion of the protocol sponsor

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2006-05; Primary Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Complete response rate

SECONDARY OUTCOMES:
Leukemia-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Bonny L. Johnson, RN, MSN — Vion Pharmaceuticals
Locations (3):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States
- Hopital Haut Leveque, Pessac, France
- University Hospital of Wales, Cardiff, Wales, United Kingdom